CLINICAL TRIAL: NCT03296358
Title: A Randomized, Double-blinded, Controlled Trial of Adding a Short Burst of Corticosteroid to the Conventional Treatment of H1 Antihistamines
Brief Title: Adding a Short Burst of Corticosteroid to the Conventional Treatment of H1 Antihistamines in Emergency Department.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 668/2017
Record Dates: First submitted 2017-09-11; First posted 2017-09-28 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Urticaria; Allergy
Keywords: Acute urticaria; Emergency department; Acute allergic syndrome; Corticosteroid; H1-Antihistamines; Chronic urticaria
MeSH Terms: conditions — Urticaria; Hypersensitivity; Emergencies; Chronic Urticaria | interventions — Dexamethasone; Calcium Dobesilate; Prednisolone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Chlorpheniramine 10 mg/amp ; 1 ampule Cetirizine 10 mg 7 tabs once daily (OD) as home medication
- Experiment 1 (Experimental): Chlorpheniramine 10 mg/amp ; 1 ampule, IV Dexamethasone 5 mg/amp; 1 ampule Cetirizine 10 mg 7 tabs 1 tab OD as home medication
  Interventions: Drug: IV Dexamethasone
- Experiment 2 (Experimental): Chlorpheniramine 10 mg/amp ; 1 ampule, IV Dexamethasone 5 mg/amp; 1 ampule Cetirizine 10 mg 7 tabs 1 tab OD as home medication Oral prednisolone 5 mg 20 tabs ; 2*2 po pc as home medication
  Interventions: Drug: IV Dexamethasone; Drug: Oral prednisolone

INTERVENTIONS:
Drug: IV Dexamethasone — The patients would be random into 3 groups. The randomization process would already be prepared into 3 groups with a number coding by the statistician who doesn't get involve in the rest of experiment. The drugs would be in the 3 group of sealed envelopes which have 3 kinds of drug combination After the envelopes are sealed, it will be code in an order of number. Experiment 1 and Experiment 2 groups would receive IV Dexamethasone in emergency department (ED).
  Other Names: Decadron; Dexasone
  Arms: Experiment 1; Experiment 2
Drug: Oral prednisolone — The patients would be random into 3 groups. The randomization process would already be prepared into 3 groups with a number coding by the statistician who doesn't get involve in the rest of experiment. The drugs would be in the 3 group of sealed envelopes which have 3 kinds of drug combination After the envelopes are sealed, it will be code in an order of number. Experiment 2 groups would receive IV Dexamethasone in ED and Oral prednisolone as home medication.
  Other Names: Orapred
  Arms: Experiment 2

SUMMARY:
A randomized, double-blinded, controlled trial of adding a short burst of corticosteroid to the conventional treatment of H1 antihistamines

DETAILED DESCRIPTION:
Research Methodology

Target Population Patients visit emergency room at King chulalongkorn memorial hospital (KCMH) age between 18-50 years who meet the following criteria of acute urticarial such as

1. eruption of wheals, central swelling of various sizes, with or without surrounding erythema; with or without angioedema
2. pruritus or occasional burning sensation
3. skin returning to normal appearance, usually within 1-24 hours

Exclusion criteria

1. patients who have urticarial for more than 48 hours
2. have severe underlying disease such as heart disease, kidney disease, liver disease
3. pregnancy
4. history of Chlorpheniramine, steroid, antihistamines allergy
5. history of antihistamine or steroid uses within 48 hours before emergency department visit
6. diabetes mellitus
7. suspected of more severe disease or severe allergic reaction
8. patients who don't have pruritus
9. patients who have history of chronic urticaria

Informed consent process The doctor who is the principal investigator or his assigned colleagues describe the research's details and methods to an enrolled patients. The documents which contain the details of the research project are also given. Inform consents then were signed before the beginning of the experiment.

The volunteer would be in a research process during their first 1-2 hours in emergency department, with the follow up time at 1 week and 1 month

After the investigator complete the inclusion and exclusion criteria, the participants would be random into 3 groups. The randomization process would already be prepared into 3 groups with a number coding by the statistician who doesn't get involve in the rest of experiment. The drugs would be in the 3 group of sealed envelopes which have 3 kinds of drug combination :

1. Control group : Chlorpheniramine 10 mg/amp ; 1 ampule and cetirizine 10 mg 7 tabs
2. Experiment group : Chlorpheniramine 10 mg/amp ; 1 ampule, Dexamethasone 5 mg/amp; 1 ampule and cetirizine 10 mg 7 tabs
3. Experiment group : Chlorpheniramine 10 mg/amp ; 1 ampule, Dexamethasone 5 mg/amp; 1 ampule, cetirizine 10 mg 7 tabs, and prednisolone 5 mg 20 tabs After the envelopes are sealed, it will be code in an order of number. All of the enrolled patients will get Chlorpheniramine 10 mg intravenous. The patients who are assigned in experiment group will get an additional Dexamethasone 5 mg intravenous. The preparation of both drugs will be result to be a 10 ml of clear fluid. The control group will get a 10 ml of sterile fluid in 10 ml syringe as a placebo. The drugs will be prepared and delivered be the nurse who knows about the research process but does not get involved in other process of the research.

After the experiment period in emergency department, all of the enrolled patients will get cetirizine 10 mg 7 tabs as a home medication. One experiment group will get prednisolone 5 mg 20 tabs. They will be appointed to an outpatient department in 1 week and 1 month for the follow up of an acute urticarial rash.

Sample size calculation Investigators do the hypothesis that the experiment groups who get both Chlorpheniramine 10 mg and Dexamethasone 5 mg intravenous would have the itch score decrease at least 2 points so this experiment wants minimal clinical difference at "2". This number got from our expert in immunology and skin disease. The standard deviation for this experiment is 2.1 from the previous research. Calculated by G*Power version 3.1 (Dusseldorf, Germany) for an independent t-test , two-tailed analysis, alpha error probability = 0.05 and power of analysis (1-beta error probability) = 0.90 The sample size for each group is 23 persons so the patients enroll in this research would be 69 persons.

Data Collection

1. Sex and age
2. Time since the first rash erupt before coming to emergency department (hrs)
3. %body surface area of rash involved
4. Urticarial activity score (UAS) before and after treatment
5. Itch score (Visual analog scale (VAS) score) by letting the patients mark a cross on a straight line. The end of the left side of a line represents "0 = no pain at all", and the end of the right side of a line represents "10 = the worst pain ever possible". The patients aren't allowed to compare the previous VAS score before doing the cross.
6. Side effect of drugs
7. Other medicine used as indicated
8. Patients' satisfaction score
9. The recurrence of rash 1 week after the rash onset
10. The recurrence of rash 1 month after the rash onset which will be evaluate by an expert in immunology and skin disease.

Data Analysis and Statistics

Descriptive statistics : Chi-square Student t-test and paired t-test for data analysis of continuous variables (such as itch score (VAS) and pair wise comparison for cumulative increase in the proportion of the "responder" over the time

Statistical significant when p-value < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Patients visit emergency room at King chulalongkorn memorial hospital (KCMH) age between 18-50 years who meet the following criteria of acute urticarial such as

  1. eruption of wheals, central swelling of various sizes, with or without surrounding erythema; with or without angioedema
  2. pruritus or occasional burning sensation
  3. skin returning to normal appearance, usually within 1-24 hours

Exclusion Criteria:

1. patients who have urticarial for more than 48 hours
2. have severe underlying disease such as heart disease, kidney disease, liver disease
3. pregnancy
4. history of chlorpheniramine maleate, steroid, antihistamines allergy
5. history of antihistamine or steroid uses within 48 hours before ED visit
6. diabetes mellitus
7. suspected of more severe disease or severe allergic reaction
8. patients who don't have pruritus
9. patients who have history of chronic urticaria

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Itch score | 60 mins
  letting the patients mark a cross on a straight line. The end of the left side of a line represents "0 = no itch at all", and the end of the right side of a line represents "10 = the worst itch ever possible". The patients aren't allowed to compare the previous VAS score before doing the cross.

SECONDARY OUTCOMES:
Chronic urticaria incidence | 1 week, 1 month
  Chronic urticaria incidence after the use of steroid compare with no steroid use in treatment.
Itch score | 0, 15, 30 mins
  letting the patients mark a cross on a straight line. The end of the left side of a line represents "0 = no itch at all", and the end of the right side of a line represents "10 = the worst itch ever possible". The patients aren't allowed to compare the previous VAS score before doing the cross.

CONTACTS AND LOCATIONS:
Overall Officials: Pakhawadee Palungwachira, M.D., Principal Investigator — King Chulalongkorn Memorial Hospital and Faculty of Medicine, Chulalongkorn University
Locations (1):
- Chulalongkorn Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided